CLINICAL TRIAL: NCT06102915
Title: Rocuronium vs Cis-atracurium: Do Rocuronium Still 'ROCKS' In Coronary Artery Bypass Grafting
Status: Completed | Type: Observational
Sponsor: Institut Jantung Negara (Other)
Responsible Party: Principal Investigator, SONG LIN LOW, Dr, Institut Jantung Negara
Other Study IDs: IJNREC/631/2023
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Neuromuscular Blockade; Postoperative Pulmonary Atelectasis; Postoperative Pulmonary Complication; Coronary Artery Disease; Coronary Artery Bypass Grafting; Hypothermic Cardiopulmonary Bypass
Keywords: Neuromuscular Blockade; Postoperative Pulmonary Atelectasis; postoperative pulmonary complication; Coronary Artery Disease; coronary artery bypass grafting; hypothermic cardiopulmonary bypass; rocuronium; cis-atracurium
MeSH Terms: conditions — Pulmonary Atelectasis; Coronary Artery Disease | interventions — Rocuronium; cisatracurium; Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rocuronium: Rocuronium 1mg/kg to be given at induction of anaesthesia and another 1mg/kg would be given when the patient is on hypothermic cardiopulmonary bypass
  Interventions: Drug: Rocuronium Bromide 10 MG/ML
- Cis-atracurium: Cis-atracurium 0.2mg/kg to be given at induction of anaesthesia and another 0.2mg/kg would be given when the patient is on hypothermic cardiopulmonary bypass
  Interventions: Drug: Nimbex 10 MG in 5 ML Injection

INTERVENTIONS:
Drug: Rocuronium Bromide 10 MG/ML — Comparative
  Other Names: Esmeron
  Groups: Rocuronium
Drug: Nimbex 10 MG in 5 ML Injection — Comparative
  Other Names: Cis-atracurium
  Groups: Cis-atracurium

SUMMARY:
The current trend in most cardiac surgeries was to use rocuronium as it provides faster recovery in train-of-four ratio compared to other aminosteroid non-depolarising neuromuscular blocker. However, as most cardiac centres' standard of care does not perform any neuromuscular monitoring nor antagonism of neuromuscular blockade effect, residual neuromuscular blockade could potentially be the key to delayed extubation. As such, Cis-atracurium's organ-independent Hofmann elimination could be in favour.

ELIGIBILITY:
Inclusion Criteria:

* All patients that undergo general anaesthesia for CABG surgery requiring neuromuscular blockade of either rocuronium or cis-atracurium

Exclusion Criteria:

1. Recent history of pulmonary infection four weeks before surgery
2. Exposed to both neuromuscular blockade within 24 hours perioperatively
3. Patients intubated or on tracheostomies pre-operatively
4. Any missing or incomplete data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that undergo general anaesthesia for CABG surgery requiring neuromuscular blockade of either rocuronium or cis-atracurium
Sampling Method: Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative pulmonary complication | 6 months
  Which neuromuscular relaxant is associated with lesser postoperative pulmonary complication

SECONDARY OUTCOMES:
Ventilation hours in ICU | 6 months
  Ventilation hours from ICU admission from OR to extubation
Requirements for Non-invasive ventilation | 6 months
  NIV duration
Incidence of postoperative atrial fibrillation | 6 months
  Incidence of postoperative atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: SONG LIN LOW, MBBS, Principal Investigator — IJN
Locations (1):
- Institut Jantung Negara, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Thomas R, Smith D, Strike P. Prospective randomised double-blind comparative study of rocuronium and pancuronium in adult patients scheduled for elective 'fast-track' cardiac surgery involving hypothermic cardiopulmonary bypass. Anaesthesia. 2003 Mar;58(3):265-71. doi: 10.1046/j.1365-2044.2003.30362.x. PMID 12638566
- [Result] Hemmerling TM, Russo G, Bracco D. Neuromuscular blockade in cardiac surgery: an update for clinicians. Ann Card Anaesth. 2008 Jul-Dec;11(2):80-90. doi: 10.4103/0971-9784.41575. PMID 18603747
- [Result] Murphy GS, Szokol JW, Vender JS, Marymont JH, Avram MJ. The use of neuromuscular blocking drugs in adult cardiac surgery: results of a national postal survey. Anesth Analg. 2002 Dec;95(6):1534-9, table of contents. doi: 10.1097/00000539-200212000-00012. PMID 12456412
- [Result] Naguib M, Samarkandi AH, Ammar A, Elfaqih SR, Al-Zahrani S, Turkistani A. Comparative clinical pharmacology of rocuronium, cisatracurium, and their combination. Anesthesiology. 1998 Nov;89(5):1116-24. doi: 10.1097/00000542-199811000-00011. PMID 9821999
- [Result] Miskovic A, Lumb AB. Postoperative pulmonary complications. Br J Anaesth. 2017 Mar 1;118(3):317-334. doi: 10.1093/bja/aex002. PMID 28186222